CLINICAL TRIAL: NCT03262051
Title: Impact of Acute and Chronic Inflammation on Cytochromes P450 Activity Measured With Dried Blood Spot
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Caroline Samer, Doctor, University Hospital, Geneva, University Hospital, Geneva
Other Study IDs: 2016-02232
Record Dates: First submitted 2017-08-21; First posted 2017-08-25 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Inflammation
Keywords: cytochromes P450; chronic inflammation; genotyping; phenotyping; acute inflammation; rheumatoid arthritis; surgery; COVID-19; SARS-CoV-2 infection
MeSH Terms: conditions — Inflammation; Arthritis, Rheumatoid; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patient with acute inflammation (surgery): patients undergoing hip surgery
  Interventions: Diagnostic Test: CYP phenotyping
- Patient with chronic inflammation: patients with rheumatoid arthritis
  Interventions: Diagnostic Test: CYP phenotyping
- Patient with acute inflammation (SARS-CoV-2 infection): patients with SARS-CoV-2 infection
  Interventions: Diagnostic Test: CYP phenotyping

INTERVENTIONS:
Diagnostic Test: CYP phenotyping — Phenotyping using a simplified version of the Geneva cocktail

SUMMARY:
Cytochromes P450, main enzymes of drug metabolism, play a prominent role in the first-pass metabolism of oral substances. Inter-individual variability in their activity due to genetic and environmental factors has been observed and may be associated with adverse therapeutic outcomes (ineffectiveness or toxicity). The inflammation, whether acute or chronic, can theoretically modulate the pharmacokinetics of drugs by modulating enzyme activity. Indeed, in vitro data and animal models, as well as more limited data in humans, indicate a down-regulation of CYP in the context of inflammation.

The cocktail approach developed and validated in Geneva ("cocktail Geneva") measures the activity of several CYP simultaneously using micro-doses of probe drugs and facilitating sampling (10uL capillary blood) on a dried blood spot.

We intend to measure the activity of CYP in an acute inflammation model (hip surgery and SARS-CoV-2 infection) and chronic inflammation (rheumatoid arthritis, RA). The effect of the biological agent tocilizumab (anti IL-6 receptor) in a treated patient subgroup (patients treated regardless of our study) will be measured after 3 months of treatment.

The main objective is to determine if interleukin 6 levels are correlated with the activity of CYP450 in patients with acute (orthopedic surgery - hip or SARS-CoV-2 infection) or chronic inflammation (RA).

Secondary objectives are:

* To correlate CYPs activities with the levels of other inflammatory markers (CRP, TNF-α, IL-1β, IFN-γ);
* To assess correlation between markers of inflammation, CYP activities and the intensity of fatigue and pain;
* To assess if tocilizumab reverse CYP activity in patients with RA after 3 months treatment;
* To assess if SARS-CoV-2 infection modify pharmacokinetic parameters of concomitant medications which are CYPs substrates

ELIGIBILITY:
--> Inclusion Criteria: For hip surgery and chronic inflammation groups

* Male and female patients diagnosed with rheumatoid arthritis or undergoing an elective hip surgery
* Age > 18 years old
* Understanding of French language and ability to give a written inform consent

For SARS-CoV-2 infection group

* Male and female patients diagnosed with SARS-CoV-2 infection (positive RT-PCR) and CRP > 30 mg/L
* Age > 18 years old
* Understanding of French language and ability to give a written inform consent

  --> Exclusion Criteria: For hip surgery and chronic inflammation groups
* Pregnant or lactating females
* Severe cardiac failure, severe edema or ascites
* Severe COPD or pulmonary embolism requiring oxygen
* Uncontrolled infection
* Active cancer
* HIV infection
* Renal impairment (defined as serum creatinine concentrations > 1.5 x ULN)
* Hepatic impairment (alteration of hepatic tests AST, ALT, bilirubin, GGT >2 x ULN)
* Inability to give blood samples
* Sensitivity to any of the drugs used
* Intake of drugs altering CYPs activity (based on [1]) except for tocilizumab

For SARS-CoV-2 infection group

* Pregnant or lactating females
* Hospitalized in intensive care unit at time of inclusion
* Hospitalized in intermediate care unit at time of inclusion
* Active cancer
* HIV infection
* Renal impairment (glomerular filtration rate < 30 mL/min/1.73m2)
* Hepatic impairment (Child-Pugh score B and C)
* Inability to give blood samples
* Sensitivity to any of the drugs used

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients included in the study will be patients with either chronic inflammation (patients with rheumatoid arthritis) or with acute inflammation (patients undergoing hip surgery or with COVID-19). All patients will be recruited at the Geneva University Hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 106 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the impact of IL6 levels on the activity of CYPs in patients with acute (post orthopaedic surgery -hip or post SARS-CoV-2 infection) and chronic (rheumatoid arthritis) inflammation. | 1 week
  The phenotyping probe drugs used in this study will be given as 2 capsules: one capsule of Omeprazole 10 mg and one capsule containing the remaining probe 'cocktail' drugs (caffeine 50 mg, flurbiprofen 10 mg, dextromethorphan 10 mg, midazolam 1 mg, bupropion 20 mg).
  The enzymatic activities of the following CYP will be assessed by specific metabolite/probe single point concentration ratios (metabolic ratios-MR) in capillary blood:
  * CYP1A2
  * CYP2B6
  * CYP2C9
  * CYP2C19
  * CYP2D6
  * CYP3A4

SECONDARY OUTCOMES:
Evaluate the correlation between the activity of CYPs and CRP levels | 1 week or 3 months
  The routine concentration of the inflammatory marker C-reactive protein (CRP) will be measured in blood
Evaluate the correlation between the activity of CYPs and TNF-α levels | 1 week or 3 months
  TNF-α blood concentrations will be measured by using the Fluorokine MAP Cytokine Multiplex Elisa.
Evaluate the correlation between the activity of CYPs and IL-1β levels | 1 week
  IL-1β blood concentrations will be measured by using the Fluorokine MAP Cytokine Multiplex Elisa.
Evaluate the correlation between the activity of CYPs and IFN-γ levels | 1 week
  IFN-γ blood concentrations will be measured by using the Fluorokine MAP Cytokine Multiplex Elisa.
Assess if tocilizumab reverse the activity of CYP in patients with RA after 3 months of treatment | 3 months
  Comparison of CYP function before and 3 months after the beginning of the Tocilizumab treatment.
Assess if SARS-CoV-2 infection modify pharmacokinetic parameters of concomitant medications which are CYPs substrates | 3 months
  Comparison of plasma concentrations of CYPs substrates, when COVID-19 patients received any CYPs substrates
Evaluate the correlation between inflammatory markers, CYP function and intensity of fatigue (MFI) and pain (NRS) | 1 week
  Function and intensity of fatigue will be measured with the validated French version of the Multidimensional Fatigue Inventory; pain will be measured with the numeric rating scale (NRS) 0 to 10 (0 = no pain and 10 = worst pain imaginable).

CONTACTS AND LOCATIONS:
Locations (1):
- Geneva University Hospitals, HUG, Geneva, Switzerland